CLINICAL TRIAL: NCT00286559
Title: Feasibility and Accuracy of Transoesophageal Harmonic Contrast Echocardiography in Assessing Myocardial Blood Flow and Blood Flow Reserve
Brief Title: Assessing Myocardial Blood Flow and Blood Flow Reserve by Transoesophageal Echocardiography (TEE)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: echo contrast agents no longer allowed in CAD patients.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 50/05
Record Dates: First submitted 2006-02-02; First posted 2006-02-03 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Coronary artery bypass graft surgery; SPECT; Adenosin
MeSH Terms: conditions — Coronary Artery Disease | interventions — contrast agent BR1; FS 069

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SonoVue
Drug: Optison

SUMMARY:
Until today it was not possible to reliably assess the function of a new bypass, i.e., to measure myocardial perfusion. Measuring intramyocardial blood flow directly after revascularisation would greatly improve the assessment of graft function. With transthoracic contrast echocardiography, myocardial perfusion can be reliably assessed, as it has been shown in numerous studies. In the first part of the study the investigators will clarify methodological aspects of contrast echocardiography. In the second part they will analyze the validity of contrast TEE in the operating room.

DETAILED DESCRIPTION:
Until today it was not possible to reliably assess the function of a new bypass, i.e., to measure myocardial perfusion. Measuring intramyocardial blood flow directly after revascularisation would greatly improve the assessment of graft function. With transthoracic contrast echocardiography myocardial perfusion can be reliably assessed, as it has been shown in numerous studies.

As there is a new transoesophageal ultrasound probe on the market which allows contrast imaging, we would like to establish contrast echocardiography in the operating room in patients undergoing CABG surgery.

Ultrasound contrast agents (e.g., SonoVue®, Optison®) consist of gas filled microspheres surrounded by a stabilizing coat. They are smaller than red blood cells and similar to blood in their rheological habit. The microspheres are injected into a peripheral or central vein. They pass lung circulation and disperse into the left heart, coronary arteries and body circulation. A few minutes after administration the low-soluble gas of the microspheres is exhaled. The interaction of the ultrasound beam with microspheres leads to oscillation of the microspheres and thereby amplification of the ultrasound signal. This technique allows enhancement of endocardial border but also visualization of myocardial perfusion and assessment of myocardial blood flow reserve. The latter requires measurement of myocardial perfusion a first time at rest and a second time during hyperemia with adenosine. The quotient of both gives myocardial flow reserve. This parameter is of paramount importance in cardiology to detect coronary artery stenosis and reduced coronary or myocardial flow reserve quantitatively.

The contrast agents as well as adenosine (a natural purine nucleoside, which can be found in all cells of the body) have a good safety profile with harmless and transient side effects. Our patients will be under anesthesia and therefore feel none of those side effects.

The study will be spread into two parts. In a first part we will clarify methodological aspects of contrast echocardiography: two different contrast agents and three different contrast imaging methods will be evaluated. One imaging method and one contrast agent will be chosen for the second part. In the second part we will analyze the validity of contrast TEE in the operating room. In addition correlation of changes in myocardial blood flow after coronary artery bypass graft (CABG) surgery and improvement in myocardial perfusion as well as global and regional function in follow-up SPECT (Single Photon Emission Computed Tomography) and transthoracic echocardiography, respectively will be evaluated. By means of these data we possibly will be able to predict success of revascularisation at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Part I: Patients with angiographically normal coronary vessels undergoing elective valve surgery or patients with coronary artery disease (CAD) who are planned for elective CABG surgery
* Part II: Patients with CAD who are planned for elective CABG surgery and who had SPECT including adenosine for hyperemia before surgery

Exclusion Criteria:

* No consent
* Acute coronary syndrome
* Acute heart failure
* Left ventricular ejection fraction < 30%
* Pronounced pulmonary artery hypertension
* Known adverse reaction against Optison or SonoVue or their components
* Severe renal or hepatic insufficiency
* Severe obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Study Completion 2008-12

PRIMARY OUTCOMES:
coronary bypass graft patency | 30 days

SECONDARY OUTCOMES:
long-term survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manfred D Seeberger, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland